CLINICAL TRIAL: NCT03261960
Title: A Safety and Efficacy Comparison of BLI4700 Bowel Preparation Versus an FDA-approved Comparator in Adult Subjects Prior to Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI4700-302
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): BLI4700 Bowel Preparation
  Interventions: Drug: BLI4700
- Control Arm (Active Comparator): FDA Approved Bowel Preparation
  Interventions: Drug: Magnesium bowel preparation

INTERVENTIONS:
Drug: BLI4700 — Oral bowel preparation
  Arms: Experimental Arm
Drug: Magnesium bowel preparation — Oral bowel preparation
  Arms: Control Arm

SUMMARY:
The objective of this study is to compare the safety and efficacy of BLI4700 bowel preparation to an FDA-approved bowel preparation as 2-day, split-dose bowel preparations prior to colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
* 18 to 85 years of age (inclusive)
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, abstinent, or vasectomized spouse).
* Negative serum pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastroparesis, gastric retention, bowel perforation, toxic colitis or megacolon.
* Subjects with ongoing severe, acute inflammatory bowel disease
* Subjects who had previous significant gastrointestinal surgeries.
* Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
* Subjects taking diuretics, anti-hypertensive medications, including angiotensin converting enzyme (ACE) inhibitors and Angiotensin II receptor blockers (ARBs), or chronic NSAIDs, that have not been stable for 30 days. NSAID use for occasional pain is not exclusionary.
* Subjects with uncontrolled hypertension (systolic blood pressure > 170 mmHg and diastolic blood pressure > 100 mmHg).
* Subjects taking antibiotics within 7 days of colonoscopy.
* Subjects with severe renal insufficiency (GFR < 30 mL/min/1.73m2).
* Subjects with known severe hepatic insufficiency (Child Pugh C)
* Subjects with cardiac insufficiency (NYHA Functional Classifications 3 or 4).
* Subjects with an abnormal and clinically significant physical examination or ECG finding at Visit 1.
* Subjects undergoing insulin therapy for any indication.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects undergoing colonoscopy for foreign body removal and/or decompression.
* Subjects who are pregnant or lactating, or intending to become pregnant during the study.
* Subjects of childbearing potential who refuse a pregnancy test.
* Subjects allergic to any preparation component.
* Subjects using drugs of abuse, including abused prescription medications.
* Subjects who are withdrawing from alcohol or benzodiazepines.
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (20):
- United States (20):
  - Braintree Research Site 119, Dothan, Alabama
  - Braintree Research Site 117, Tucson, Arizona
  - Braintree Research Site 108, Little Rock, Arkansas
  - Braintree Research Site 110, Little Rock, Arkansas
  - Braintree Research Site 139, Palmetto Bay, Florida
  - Braintree Research Site 124, Oak Lawn, Illinois
  - Braintree Research Site 134, Indianapolis, Indiana
  - Braintree Research Site 112, Chevy Chase, Maryland
  - Braintree Research Site 141, Towson, Maryland
  - Braintree Research Site 125, Chesterfield, Missouri
  - Braintree Research Site 102, St Louis, Missouri
  - Braintree Research Site 145, Egg Harbor, New Jersey
  - Braintree Research Site 114, Poughkeepsie, New York
  - Braintree Research Site 105, Asheville, North Carolina
  - Braintree Research Site 115, Charlotte, North Carolina
  - Braintree Research Site 137, Raleigh, North Carolina
  - Braintree Research Site 101, Raleigh, North Carolina
  - Braintree Research Site 107, Greenville, South Carolina
  - Braintree Research Site 131, Charlottesville, Virginia
  - Braintree Research Site 121, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm | Control Arm
Started (Safety population - all patients that took preparation.) | 190 | 199
Completed | 176 | 185
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Population: Safety population - all patients that took preparation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Control Arm | Total
Number analyzed (Participants) | 190 | 199 | 389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 152 | 280
  >=65 years | 62 | 47 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.2) | 57.3 (10.8) | 57.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 113 | 225
  Male | 78 | 86 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 16 | 35
  Not Hispanic or Latino | 171 | 183 | 354
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 11 | 19
  White | 177 | 183 | 360
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 190 | 199 | 389
Renal Insufficiency (GFR < 60) [Count of Participants; unit: Participants] — Subjects with baseline GFR < 60 mL/min/1.73 m2
  Participants | 16 | 14 | 30
Diabetic [Count of Participants; unit: Participants] — Subjects with a medical history of diabetes
  Participants | 20 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With Successful Bowel Cleansing
Description: % of subjects with successful bowel preparation rated by colonoscopist on a 4 point scale (1=poor to 4=excellent)
Time Frame: Day of colonoscopy
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 190 | 198
Participants | 175 | 174
Statistical Analysis 1: Comparison: Experimental Arm vs Control Arm; Test type: Non-Inferiority — Non-inferiority margin was set at 10%; p < 0.001, Cochran-Mantel-Haenszel

2. Other Pre Specified Outcome: Abdominal Pain (Solicited Reports)
Description: Percentage of patients who reported abdominal pain (with associated severity) when directly queried by study personnel, out of all patients that reported that event.
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 190 | 199
percentage of patients
  Mild | 82 | 100
  Moderate | 16 | 0
  Severe | 2 | 0

3. Other Pre Specified Outcome: Abdominal Distension (Solicited Reports)
Description: Percentage of patients who reported abdominal distension (with associated severity) when directly queried by study personnel, out of all patients that reported that event.
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 190 | 199
percentage of patients
  Mild | 73 | 69
  Moderate | 27 | 31
  Severe | 0 | 0

4. Other Pre Specified Outcome: Nausea (Solicited Reports)
Description: Percentage of patients who reported nausea (with associated severity) when directly queried by study personnel, out of all patients that reported that event.
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 190 | 199
percentage of patients
  Mild | 74 | 94
  Moderate | 20 | 6
  Severe | 6 | 0

5. Other Pre Specified Outcome: Vomiting (Solicited Reports)
Description: Percentage of patients who reported vomiting (with associated severity) when directly queried by study personnel, out of all patients that reported that event.
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 190 | 199
percentage of patients
  Mild | 53 | 33
  Moderate | 47 | 67
  Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Experimental Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/199
Serious Adverse Events (participants affected / at risk) | 0/190 | 1/199
Other Adverse Events (participants affected / at risk) | 5/190 | 2/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=190) | Control Arm (N=199)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=190) | Control Arm (N=199)
Liver function test increased (Investigations) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT03261960/Prot_SAP_000.pdf